CLINICAL TRIAL: NCT06975189
Title: Lung Ultrasound to Reduce the Number of Chest X-rays in Very Preterm Infants in the First 2 Weeks After Birth: A Randomised Controlled Trial
Brief Title: MINImising Total Radiation EXposure in Preterm Infants
Acronym: MINI T-Rex
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Western Health, Australia (Other Government)
Responsible Party: Principal Investigator, Arun Sett, Neonatologist, Western Health, Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 115953
Record Dates: First submitted 2025-04-09; First posted 2025-05-16 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Neonatal Respiratory Distress Syndrome; PreTerm Neonate
Keywords: Lung ultrasound; Respiratory Distress Syndrome; Prematurity
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinicians and participants will be unblinded to the study intervention. All outcome analysis will be performed blinded to the study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lung ultrasound group (Experimental): Infants randomised to this group will have lung ultrasound as their first
  Interventions: Device: Lung ultrasound group
- Standard care (Active Comparator): Infants in the standard arm will receive chest X-ray as their first form of lung imaging. Lung ultrasound will not be permitted in this group.
  Interventions: Diagnostic Test: Standard Care

INTERVENTIONS:
Device: Lung ultrasound group — Infants in the intervention arm will receive lung ultrasound as their first line imaging. Clinicians will be permitted to order a chest x-ray if they require further information or if the lung ultrasound findings are inconclusive or not consistent with the clinical findings.
  Arms: Lung ultrasound group
Diagnostic Test: Standard Care — Infants in the standard group will receive chest X-ray as their first line imaging tool. Lung ultrasound will not be permitted in this group.
  Arms: Standard care

SUMMARY:
Being born too early (preterm birth) is the leading cause of death in children world-wide. In Australia, 97% of very preterm babies who are admitted to Neonatal Intensive Care Units need breathing support after birth to survive. Despite this significant global impact, neonatal clinicians have few tools available to guide breathing support. Currently, the only lung imaging tool that is routinely used in the Neonatal Intensive Care Unit is a chest X-ray. To reduce radiation exposure, chest X-rays are usually only performed one or two times a day. As chronic lung disease in babies who survive preterm birth is increasing, there is an urgent need to develop new ways to monitor the lungs of these fragile babies.

Lung ultrasound is a form of imaging that is fast, gentle and radiation free. However, it has not been routinely adopted into caring for preterm babies in most countries. This is because there are no randomised controlled trials that have demonstrated the benefit and safety of using lung ultrasound as the first-line imaging tool in preterm babies. The investigators will conduct a randomised controlled trial to demonstrate that lung ultrasound is a quick, safe and accurate alternative to chest x-rays in preterm babies.

DETAILED DESCRIPTION:
Preterm babies are born with underdeveloped, fragile lungs and commonly develop respiratory distress syndrome. In Australia, 97% of preterm babies who are admitted to Neonatal Intensive Care Units need breathing support after birth. Respiratory support is vital to keep babies alive but is associated with short- and long-term lung damage. Unfortunately, many babies who survive preterm birth develop bronchopulmonary dysplasia (BPD), leading to poor health outcomes in adulthood.(2) Despite years of research, chronic lung disease is increasing.

Clearly, it is critical that clinicians have effective tools to guide breathing support. Currently, the only lung imaging tool that is routinely used in the Neonatal Intensive Care Unit is chest X-ray (CXR). The fundamental principle of use of ionising radiation in any population is to limit radiation exposure to as low as reasonably achievable (ALARA). To achieve this currently, the use of CXR is usually limited to once or twice a day. In addition CXR are performed by a specialised technician and are not always immediately available, delaying the time to diagnosis. Given the rapid and unpredictable changes in a preterm baby's lung disease, reliance on repeated CXR is fraught with risk. There is an urgent need to develop reliable tools that provides real-time and accurate feedback to guide breathing support in preterm babies.

New monitoring tools should be safe and improve outcomes. Lung ultrasound is a gentle form of lung imaging that is ideally suited for preterm babies. It is radiation free, readily available and does not require excessive handling of the baby. Ultrasound is already routinely used to image the brain and hearts of preterm babies and systems are available in all Neonatal Intensive Care Units in Australia. Several observational studies have demonstrated that lung ultrasound is accurate in diagnosing common neonatal respiratory disorders including pneumothorax, respiratory distress syndrome, transient tachypnoea of the newborn and the need for mechanical ventilation. Not all features of lung ultrasound are interchangeable with CXR measures of lung aeration in preterm infants. Lung ultrasound has a stronger relationship with an infant's respiratory support requirements than CXR. Only one study to date has assessed the ability of lung ultrasound to guide surfactant replacement in a randomized setting. Despite the growing body of evidence that lung ultrasound may be a suitable alternative to CXR, it has not been routinely adopted into clinical practice. This is because no randomized controlled trial has assessed the benefit and safety of using lung ultrasound as the first-line imaging tool in preterm babies. Furthermore, despite no evidence of benefit, some centres have already implemented lung ultrasound into routine practice. Before lung ultrasound can be widely implemented in preterm babies, it must be demonstrated to be beneficial and safe.

The investigators hypothesise that in preterm babies born <32 weeks' gestation, lung ultrasound will significantly reduce radiation exposure and be a safe alternative to CXR. This will be addressed by conducting an open label, randomised controlled trial at Joan Kirner Women's and Children's, Sunshine Hospital, Victoria.

The primary aim of this study is to evaluate whether the use of lung ultrasound as the primary lung imaging modality in preterm babies born <32 weeks' gestation reduces radiation burden.

Secondary aims include assessment of the safety and acceptability of lung ultrasound as the first line imaging tool, and additional signals of benefit including time to receive lung imaging and initiation of treatment, and duration of breathing support. To assess safety, the investigators will report the rate of key protocol defined adverse and serious adverse events in the intervention and control groups. Feasibility will be determined by protocol defined criteria for operational and clinical feasibility. Cost effectiveness will be determined by reporting the microcosts of each imaging tool and comparing the differential costs between the lung ultrasound and chest X-ray. Finally, the investigators will assess the acceptability to neonatal healthcare workers of lung ultrasound as the first-line imaging tool.

ELIGIBILITY:
Inclusion Criteria:

All infants born <32 weeks' gestation and admitted to the neonatal intensive care unit (NICU) who require lung imaging for respiratory indications will be considered eligible. Each infant must meet all the following criteria to be enrolled in this study:

* The infant is born from 22 to 31+6 weeks' gestation by best obstetric estimate and admitted to the NICU
* The infant is considered to require lung imaging for respiratory indications
* The infant has a parent/guardian who can provide informed consent.

Exclusion Criteria

* The infant will only require CXR to be performed solely to confirm device position i.e. central line, endotracheal tube, gastric tubes
* The infant will only require CXR to be performed for specifically for non-respiratory indications i.e. assessment of cardiac silhouette
* The infant's Clinician has concern regarding clinical stability and tolerability of ultrasound scans
* The infant's skin integrity will not tolerate ultrasound gel
* Refusal of informed consent by their parent/guardian/legally acceptable representative
* The infant does not have a parent/guardian who can provide informed consent.

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
The mean difference in number of x-rays and radiation exposure in the intervention group | Until day 14 of life
  The total number of chest X-rays performed in the study period

SECONDARY OUTCOMES:
The mean difference of X-rays for entire admission (until discharge or death) | From date of randomization until the date of discharge or date of death from any cause, whichever came first, assessed up to 12 months
  Total number of x-rays performed from enrolment in study until death or discharge from hospital
The mean difference of X-rays and radiation exposure by gestational age at birth | Until day 14 of life
  The total number of CXR performed in the study period stratified by gestational groups (< 28 weeks' gestation and >/= to 28 weeks' gestation)
Time to administering surfactant if clinically indicated | Until day 14 of life
  The mean difference in minutes to administer surfactant if clinically indicted between the lung ultrasound and chest x-ray groups
Proportion of infants in the intervention arm who require CXR as first-line imaging due to lung ultrasound not being available | Until day 14 of life
  The number of CXRs performed after a lung ultrasound is performed in the intervention group due to the ultrasound clinicians or system not being available.
Cost-effectiveness | Until day 14 of life
  The differential costs between the intervention and control groups determine from a time-in-motion analysis of a pre-determined sub sample of the study population (n=10 patients per group)

OTHER OUTCOMES:
Serious adverse event [1] | During or within 1 hour after each scheduled lung imaging assessment
  Oxygen requirement of fraction of inspired oxygen (FiO2) ≥20% of baseline for 2 hours or more after the lung imaging assessment
Serious adverse event [2] | During or within 1 hour after each scheduled lung imaging assessment
  Acute oxygen desaturation (peripheral oxygen saturations [SpO2] <90%) that required the lung imaging to be terminated
Serious adverse event [3] | During or within 1 hour after each scheduled lung imaging assessment
  Requirement of escalation of respiratory support
Serious adverse event [4] | During or within 1 hour after each scheduled lung imaging assessment
  Apnoea requiring stimulation or other intervention that required the lung imaging to be terminated
Serious adverse event [5] | Within 1 hours of each scheduled lung imaging assessment a photograph of the area will be taken and blindly scored using Hume-T scoring system
  For infants born <24 weeks' gestation, breech of skin integrity or skin irritation associated with lung imaging within 1 hour of imaging episode
Serious adverse event [6] | From the date of randomisation until 14 days
  Allocated imaging not being available and alternative imaging required
Adverse event [1] | During or within 24 hours after each scheduled lung imaging assessment
  Any death
Adverse event [2] | During or within 24 hours after each scheduled lung imaging assessment
  Pulmonary haemorrhage
Adverse event [3] | During or within 24 hours after each scheduled lung imaging assessment
  Administration of epinephrine or use of chest compressions
Adverse event [4] | During or within 1 hour after each scheduled lung imaging assessment
  Unplanned extubation
Adverse event [5] | Within first 2 weeks of age
  In the intervention group, a significant delay in diagnosis and initiation of appropriate intervention for the following conditions due to lung ultrasound being inconclusive and a CXR being required to confirm diagnosis as determined by the clinical team:
  * Significant pneumothorax
  * Significant pleural effusion
  * Severe respiratory distress syndrome requiring surfactant replacement therapy
Duration and level of mechanical ventilation and/or other respiratory support | From date of randomisation until death or discharge, whichever comes first, maximum 12 months
  Days of supplemental oxygen
Duration of invasive and non invasive ventilation | From date of randomisation until death or discharge, whichever comes first, maximum 12 months
  Days of respiratory support including mechanical ventilation, continuous positive airway pressure and nasal high flow therapy
Post natal corticosteroid use | From date of randomisation until death or discharge, whichever comes first, maximum 12 months
  Use of postnatal steroids, including types, timing and accumulated doses
Incidence of Air leak | From date of randomisation until death or 2 weeks of age, whichever comes first, 2 weeks
  Incidence of pulmonary interstitial emphysema or pneumothorax
Use of Volume expansion (crystalloid or colloid) | From date of randomisation until death or 2 weeks of age, whichever comes first, 2 weeks
  Total amount of volume expansion (in ml/kg) given during study duration
Use of inotropic support | From date of randomisation until death or 2 weeks of age, whichever comes first, 2 weeks
  Maximum level of inotropic support given (drug and dose) during study duration
Blood transfusion administration | From date of randomisation until death or 2 weeks of age, whichever comes first, 2 weeks
  Total blood transfused in ml/kg during study duration
Incidence of patent ductus arteriosus | From date of randomisation until death or 2 weeks of age, whichever comes first, 2 weeks
  Incidence of patent ductus arteriosus requiring medical or surgical treatment during study duration
Incidence of retinopathy of prematurity | From date of randomisation until death or discharge, whichever comes first, maximum 6 months
  Incidence of retinopathy of prematurity stratified by grade
Incidence of necrotising enterocolitis | From date of randomisation until death or 2 weeks of age, whichever comes first, 2 weeks
  Incidence of Stage 2 or higher necrotising enterocolitis for study duration
Incidence of intraventricular haemorrhage (IVH) | From date of randomisation until death or discharge, whichever comes first, maximum 6 months
  Incidence of IVH over entire admission
Incidence of periventricular leukomalacia (PVL) | From date of randomisation until death or discharge, whichever comes first, maximum 12 months
  Incidence of PVL during entire admission
Duration of admission | From date of randomisation until death or discharge, whichever comes first, maximum 12 months
  Duration of entire hospital admission u
Diagnosis of BPD at 36 weeks | From date of randomisation until death or discharge or 36 weeks post menstrual age, whichever comes first, maximum 36 weeks
  BPD status at 36 weeks defined by the standard oxygen reduction (ORT) test
Death | From date of randomisation until death or discharge or 36 weeks post menstrual age, whichever comes first, maximum 6 months
  Survival status/date of death during hospital stay / cause and location of death

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data will be shared to research parties who have a sound research proposal and prior institutional review board approval.